CLINICAL TRIAL: NCT04792307
Title: Feasibility RCT of Neuromuscular Electrical Stimulation; an Intervention to Maintain and Improve neuroMuscular Function During Periods of Immobility
Brief Title: Neuromuscular Electrical Stimulation Study
Acronym: IMMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20HC006
Record Dates: First submitted 2021-02-09; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Sarcopenia
Keywords: Frailty,; Immobility; Electrical Stimulation; High protein
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Intervention Model Description: will randomly allocate participants offering half of them additional protein supplementation over and above their ordinary diet
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular electrical stimulation (NMES) to one leg (Other): * NMES left leg, no high protein ice cream supplementation
  * NMES right leg, no high protein ice cream supplementation
  Interventions: Other: Neuromuscular electrical stimulation , no high protein ice cream supplementation
- High protein ice cream supplementation (Other): * NMES left leg, high protein ice cream supplementation
  * NMES right leg, high protein ice cream supplementation
  Interventions: Other: Neuromuscular electrical stimulation , no high protein ice cream supplementation

INTERVENTIONS:
Other: Neuromuscular electrical stimulation , no high protein ice cream supplementation — A trained operator applies Neuromuscular electrical stimulation treatment to one leg, for approximately 30 minutes per session, three sessions per week with or without high protein ice cream. Treatment can stimulate the nerve controlling the vastus lateralis muscle in the thigh or the nerve controlling the tibialis anterior muscle in the lower leg, or both. In our study, we will aim to stimulate both nerves and muscle groups, on the basis that the maximal effect with result from the maximal amount of muscle stimulated.Treatment is adjusted to generate a specific force and maintained for up to 5 minutes, followed by a rest period and then repeated three times over the typical 30-minute session. The stimulation can vary according to the frequency (pulses per second, typically 10-50Hz).
  Additional protein supplementation: high protein ice cream :a single doses of a high protein supplement after each bout of neuromuscular electrical stimulation,
  Other Names: Neuromuscular electrical stimulation with high protein ice cream supplementation

SUMMARY:
In this study, the investigators will use feasibility RCT design to determine whether it is justifiable to conduct a large-scale clinical trial of neuromuscular electrical stimulation with or without additional protein supplementation in hospitalised patients who are temporarily immobilised following a fragility fracture. Muscle thickness, muscle strength, patients' mobility and self-care will be assessed at baseline and after 6-wk trial duration or until patients discharged from hospital. Outcomes will include participants' recruitment rate, tolerability and accessibility and their characteristics.

DETAILED DESCRIPTION:
In frail elderly people with existing sarcopenia, muscle mass, muscle strength and muscle function during immobility after lower limb fractures are impaired and affect their functional abilities to achieve activities of daily living. To reverse these consequences, limited intervention studies show that resistance exercise training and protein supplement at least partly reverses sarcopenia. However, guidelines do not currently advise specific protein supplementation as a treatment to prevent or reverse sarcopenia. Additionally, these exercises are difficult to perform in adequate intensity when patients are ill, tired, or in pain and these same factors may reduce appetite. In this study, the investigators aim to evaluate the effect of neuromuscular electrical stimulation with and without a high protein oral nutritional supplement.

Methods:

In this study, the investigators will use feasibility RCT design to determine whether it is justifiable to conduct a large-scale clinical trial of neuromuscular electrical stimulation with or without additional protein supplementation in hospitalised patients who are temporarily immobilised following a fragility fracture. Muscle thickness, muscle strength, patients' mobility and self-care will be assessed at baseline and after 6-wk trial duration or until patients discharged from hospital. Outcomes will include participants' recruitment rate, tolerability and accessibility and their characteristics.

Discussion This study addresses the effects of neuromuscular electrical stimulation with or without high protein supplements on mobility, self-care, muscle mass and strength in immobile older people with frailty after lower limb fracture. The information from this study may justify a large-scale clinical trial of using electrical stimulation with or without high protein supplement.

ELIGIBILITY:
Inclusion Criteria:

* >/=65 years
* Hospitalised due to incident fragility fracture (hip, spine, pelvis, rib, upper limb, lower limb)
* Immobile 72 hours after admission or completion of surgery whichever is the later.
* Predicted date of discharge >/= 7 days after recruitment

Exclusion Criteria:

* Unable to give valid informed consent

  * Residence outside catchment area of hospital (likely to be moved during the study period)
  * Unable to communicate in English sufficiently to participate in neuromuscular electrical stimulation.
  * Implanted medical device (e.g. pacemaker)
  * Any other contraindications to neuromuscular electrical stimulation (e.g. injury to the stimulation sites)
  * Leg amputation or any pre-injury conditions affecting a leg unilaterally such as hemiparesis
  * Dysphagia for liquids
  * Protein supplementation clinically indicated and prescribed
  * End stage renal failure
  * Obesity (BMI>30)
  * End of life, for any reason
  * Any other clinical reason why rehabilitation is not clinically indicated
  * Within 10 days of being symptom free having been COVID-19 positive (PCR testing or clinical criteria), or other barrier nursed patients
  * Lactose intolerance

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Lower limb muscle strength | "Change from Baseline lower limb muscle strength at 6 weeks"
  using A hand-held dynamometer for both vastus lateralis and tibialis anterior muscles
Hand grip strength | "Change from Baseline Hand grip strength at 6 weeks"
  using a standard device
Ultrasound | "Change from Baseline lower limb muscle thickness at 6 weeks"
  Ultrasound parameters of vastus lateralis and tibialis anterior muscles (thickness, pennation angle, echogenicity).
iEMG derived motor unit structure and function | "Change from Baseline lower limb muscle control at 6 weeks"
  intramuscular electromyography (iEMG) measures of muscle control
Elderly Mobility Scale | "Change from Baseline functional independence at 6 weeks"and " 6 months"
  measuring 9 domains from very fit 1 to terminally ill 9
Nottingham Extended ADL | "Change from Baseline functional independence at 6 weeks"and " 6 months"
  The Answers to the questions should be given whenever possible by the person who is the subject of the questionnaire Answers should be recorded by ticking one box for each question
Disability and functional independence using Barthel ADL score. | Change from Baseline functional independence at 6 weeks "and " 6 months"]
  an ordinal scale used to measure performance in activities of daily living (ADL). variables describing ADL and mobility are scored, a higher number being a reflection of greater ability to function independently following hospital discharge.

SECONDARY OUTCOMES:
Tolerability measurement | "up to 6 weeks"
  high number yes, low number no
Pain/Visual analogue scores | "Change from Baseline functional independence at 6 weeks "
  1 less pain, 10 severe pain
Mortality Rate | At 6 months after recruitment
  the number of participants who died within 6 months period after recruitment.
Number of protein supplementation doses consumed | "up to 6 weeks"
  How many cups participants consumed 1 cup lowest and 18 cups highest
Acceptability verbal questionnaire of Neuromuscular stimulation | "up to 6 weeks"
  yes / no answers, number of sessions participants say yes they accept or no not accept
Number of treatment sessions of Neuromuscular stimulation | "up to 6 weeks"
  number of treatment sessions 1 lowest and 18 highest
Duration of treatment sessions of Neuromuscular stimulation | "up to 6 weeks"
  number of weeks participants received Neuromuscular stimulation 1 week lowest, 6 weeks highest

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kofali, Study Chair — Nottingham University Hospitals NHS Trust

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) available only to those involved in the research project

REFERENCES:
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Background] Wilkinson DJ, Piasecki M, Atherton PJ. The age-related loss of skeletal muscle mass and function: Measurement and physiology of muscle fibre atrophy and muscle fibre loss in humans. Ageing Res Rev. 2018 Nov;47:123-132. doi: 10.1016/j.arr.2018.07.005. Epub 2018 Jul 23. PMID 30048806
- [Background] Rudrappa SS, Wilkinson DJ, Greenhaff PL, Smith K, Idris I, Atherton PJ. Human Skeletal Muscle Disuse Atrophy: Effects on Muscle Protein Synthesis, Breakdown, and Insulin Resistance-A Qualitative Review. Front Physiol. 2016 Aug 25;7:361. doi: 10.3389/fphys.2016.00361. eCollection 2016. PMID 27610086
- [Background] Anthony K, Robinson K, Logan P, Gordon AL, Harwood RH, Masud T. Chair-based exercises for frail older people: a systematic review. Biomed Res Int. 2013;2013:309506. doi: 10.1155/2013/309506. Epub 2013 Sep 9. PMID 24089670
- [Background] Welch C, Majid Z, Greig C, Gladman J, Masud T, Jackson T. Interventions to ameliorate reductions in muscle quantity and function in hospitalised older adults: a systematic review towards acute sarcopenia treatment. Age Ageing. 2021 Feb 26;50(2):394-404. doi: 10.1093/ageing/afaa209. PMID 33098419
- [Background] Dacombe PJ, Clement RGE, Woodard J, Sahota O. Poor nutritional intake in acute fractured neck of femur admission - is this well described clinical problem still under-managed? International Journal of Surgery (Abtracts) 2010 : 8 ; 501-578
- [Background] Jones S, Man WD, Gao W, Higginson IJ, Wilcock A, Maddocks M. Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2016 Oct 17;10(10):CD009419. doi: 10.1002/14651858.CD009419.pub3. PMID 27748503
- [Background] Symons TB, Sheffield-Moore M, Wolfe RR, Paddon-Jones D. A moderate serving of high-quality protein maximally stimulates skeletal muscle protein synthesis in young and elderly subjects. J Am Diet Assoc. 2009 Sep;109(9):1582-6. doi: 10.1016/j.jada.2009.06.369. PMID 19699838
- [Background] Martin HJ, Yule V, Syddall HE, Dennison EM, Cooper C, Aihie Sayer A. Is hand-held dynamometry useful for the measurement of quadriceps strength in older people? A comparison with the gold standard Bodex dynamometry. Gerontology. 2006;52(3):154-9. doi: 10.1159/000091824. PMID 16645295
- [Background] Lunt E, Ong T, Gordon AL, Greenhaff PL, Gladman JRF. The clinical usefulness of muscle mass and strength measures in older people: a systematic review. Age Ageing. 2021 Jan 8;50(1):88-95. doi: 10.1093/ageing/afaa123. PMID 32706848
- [Background] Tarquinio C, Kivits J, Minary L, Coste J, Alla F. Evaluating complex interventions: perspectives and issues for health behaviour change interventions. Psychol Health. 2015 Jan;30(1):35-51. doi: 10.1080/08870446.2014.953530. Epub 2014 Oct 21. PMID 25140439
- [Background] Collin C, Wade DT, Davies S, Horne V. The Barthel ADL Index: a reliability study. Int Disabil Stud. 1988;10(2):61-3. doi: 10.3109/09638288809164103. PMID 3403500
- [Background] Gladman JR, Lincoln NB, Adams SA. Use of the extended ADL scale with stroke patients. Age Ageing. 1993 Nov;22(6):419-24. doi: 10.1093/ageing/22.6.419. PMID 8310887
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Stratton RJ, Hackston A, Longmore D, Dixon R, Price S, Stroud M, King C, Elia M. Malnutrition in hospital outpatients and inpatients: prevalence, concurrent validity and ease of use of the 'malnutrition universal screening tool' ('MUST') for adults. Br J Nutr. 2004 Nov;92(5):799-808. doi: 10.1079/bjn20041258. PMID 15533269
- [Background] Laufer Y, Shtraker H, Elboim Gabyzon M. The effects of exercise and neuromuscular electrical stimulation in subjects with knee osteoarthritis: a 3-month follow-up study. Clin Interv Aging. 2014 Jul 17;9:1153-61. doi: 10.2147/CIA.S64104. eCollection 2014. PMID 25083133
- [Background] Asakawa Y, Jung JH, Koh SE. Neuromuscular electrical stimulation improves strength, pain and weight distribution on patients with knee instability post surgery. Physical therapy rehabilitation science. 2014;3(2):112-8.
- [Background] Chen RC, Li XY, Guan LL, Guo BP, Wu WL, Zhou ZQ, Huo YT, Chen X, Zhou LQ. Effectiveness of neuromuscular electrical stimulation for the rehabilitation of moderate-to-severe COPD: a meta-analysis. Int J Chron Obstruct Pulmon Dis. 2016 Nov 28;11:2965-2975. doi: 10.2147/COPD.S120555. eCollection 2016. PMID 27932876